CLINICAL TRIAL: NCT07088172
Title: Clinical Effects of Keratinized Mucosa Augmentation Around Dental Implant With Free Gingival Graft in Different Surgical Timing at Mandibular Posterior Sites
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-064
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Edentulous Alveolar Ridge In Mandible

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- free gingival grafting during the second stage of implant surgery (Experimental): Free gingival graft surgery performed simultaneously with the second stage of the implant surgery, followed by the restoration 6-8 weeks later.
  Interventions: Procedure: free gingival grafts during the second stage of implant surgery
- free gingival grafts prior to the implantation (Other): Free gingival graft surgery is performed 6-8 weeks before implant placement
  Interventions: Procedure: free gingival grafts prior to the implantaion

INTERVENTIONS:
Procedure: free gingival grafts during the second stage of implant surgery — Free gingival graft surgery performed simultaneously with implant stage II, followed by upper restoration 6-8 weeks later.
  Arms: free gingival grafting during the second stage of implant surgery
Procedure: free gingival grafts prior to the implantaion — Free gingival graft surgery performed 6-8 weeks before implant placement
  Arms: free gingival grafts prior to the implantation

SUMMARY:
This study aims to compare clinical outcomes and tissue stability at implant sites in the mandibular posterior region with insufficient buccal keratinized gingiva. It will assess the use of free gingival grafts either before or during the second stage of implant surgery.

DETAILED DESCRIPTION:
To compare the clinical outcomes and the differences in hard and soft tissue stability at implant sites with insufficient buccal keratinized gingiva in the mandibular posterior region, where free gingival grafts are applied either before implant surgery or concurrently during the second stage of implant surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, gender unrestricted;
* partially edentulous in the mandible posterior area, planned for implant-supported fixed restoration;
* Buccal keratinized mucosa width at the implant site is less than 2mm, with the transplantation area not exceeding 2 teeth;
* No soft tissue augmentation performed at the site prior to surgery;
* Overall health is good, with no systemic diseases that may affect bone metabolism or wound healing;
* Good periodontal condition, no progressive alveolar bone resorption, no periodontal abscess;
* Smoking ≤ 10 cigarettes per day.

Exclusion Criteria:

* Uncontrolled metabolic diseases;
* Severe periodontal disease, with unstable periodontal condition;
* Smoking > 10 cigarettes per day;
* Unwilling to participate in the follow-up of this study;
* Other conditions that do not meet the requirements for implant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Width of Keratinized Mucosa, KMW | Preoperative\Immediate postoperative\2 months postoperative\6 months postoperative

SECONDARY OUTCOMES:
Thickness of Keratinized Mucosa, KMT | Preoperative\ Immediate postoperative\2 months postoperative\6 months postoperative
Postoperative Discomfort | follow-up time point(at least 6 months after restoration)
  Visual Analog Scale
Plaque Index,PI | follow-up time point(at least 6 months after restoration)
Bleeding on Probing, BOP | follow-up time point(at least 6 months after restoration)
Peri-implant Probing Depth, PPD | follow-up time point(at least 6 months after restoration)
Marginal Bone Loss, MBL | follow-up time point(at least 6 months after restoration)
Patient Satisfaction | follow-up time point(at least 6 months after restoration)
  Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- The Stomatology Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China